CLINICAL TRIAL: NCT00929825
Title: Effects of Mechanical and Electrical Sialogogues in Stimulation of the Flow and Biochemical Composition of Saliva in Patients Transplanted With Hematopoietic Stem Cells
Brief Title: Therapies for Salivary Flux Stimulation in Patients Transplanted With Hematopoietic Stem Cells
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The Hospital had the Unit of Stem cells Tranplantion suspended
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Tania Mara Pimenta Amaral (Unknown)
Responsible Party: Principal Investigator, Tarcilia Aparecida da Silva, Associate Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 0520; Not aplicable
Record Dates: First submitted 2009-06-04; First posted 2009-06-30 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Mucositis
Keywords: Salivary stimulation; Transplantation of hematopoietic stem cells; Hyperboloid; Transcutaneous Electrical Stimulation
MeSH Terms: conditions — Mucositis | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Elastomers (Experimental): Patients will use hyperboloid as mechanical salivary stimuli. Patients will chew hyperboloid 3 times a day
  Interventions: Device: mechanical stimulation (Elastomers)
- TENS (Experimental): TENS is a eletric stimuli that will be use in the skin near to parotid glands. Patients will receive TENS treatment as eletric salivary stimuli. Patients will receive TENS stimuli once a day for 15 days
  Interventions: Procedure: TENS
- Elastomers+TENS (Experimental): Patients will receive TENS plus hyperboloid as eletric and mechanical treatment for salivary stimuli
  Interventions: Device: mechanical stimulation (Elastomers); Procedure: TENS
- No therapy (control) (No Intervention): Patients will not receive intervention

INTERVENTIONS:
Device: mechanical stimulation (Elastomers) — The instrument of mastication, sialogogue should be used 4 times a day for 10 minutes each time always after meals
  Arms: Elastomers; Elastomers+TENS
Procedure: TENS — transcutaneous electrical stimulation
  Arms: Elastomers+TENS; TENS

SUMMARY:
The transplantation of hematopoietic stem cells (THSC) is a therapeutic modality developed for the treatment of various diseases such as leukemia, bone marrow aplasia, lymphomas, multiple myeloma, among others. Most patients who undergo the THSC usually have oral manifestations as a result of immunosuppression achieved by chemotherapy and/or radiotherapy. The most common complications are the reduction of salivary flow, mucositis and graft-versus-host disease (GVHD). These conditions can be very debilitating and interfere with medical therapy, leading to systemic complications, affecting the prognosis and increasing the length of hospitalization of the patient and the costs of treatment. To date, there is no protocol that prevents the reduction of salivary flow and minimizes the occurrence of mucositis and GVHD in these patients. This study aims to verify the effectiveness of treatment with two sialogogues (Hyperboloid and TENS [transcutaneous electrical stimulation]) to restore the flow and biochemical composition of saliva in patients undergoing THSC myeloablative and non-myeloablative conditionating regime.

DETAILED DESCRIPTION:
It will be included in the sample a total of 60 patients undergoing hematopoietic stem cell transplantation (THSC) at the Clinical Hospital. Patients will be randomly divided into four groups, each with 15 subjects: group I patients who will use only the mechanical sialogogue; group II patients who will make use of electrical sialogogue (TENS); group III patients who will make use of mechanical sialogogue associated with TENS and group IV patients who will not receive therapy (control).

The project will present the following experimental design:

1. Selection of patients to be subjected to the transplantation of hematopoietic stem cells;
2. Implementation of a reference sialometry;
3. Institution of therapy with mechanical and electrical sialogogue;
4. Clinical examination, assessment of the occurrence of mucositis and obtention of saliva samples pre- and post-THSC;
5. Qualitative analysis of saliva (turbidity, viscosity and color);
6. Biochemical analysis of saliva;
7. Statistical analysis of data.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to THSC at Clinical Hospital of Federal University who underwent a myeloablative or a non-myeloablative conditioning regime
* Age over 16 years
* Oral mucosa intact on the first day of conditioning
* Ability to cooperate with treatment

Exclusion Criteria:

* Cases with no clinical follow up
* Patients who refuse to participate
* Patients with no ability to cooperate with treatment

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Salivary flux | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Tarcilia A Silva, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Faculty of Dentistry of Federal University of Minas Gerais, Belo Horizonte, Minas Gerais/Belo Horizonte, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Oral Surg Oral Med Oral Pathol Oral Radiol. 2012 May;113(5):628-37. doi: 10.1016/j.oooo.2011.10.012. Epub 2012 Apr 12.
  Effect of salivary stimulation therapies on salivary flow and chemotherapy-induced mucositis: a preliminary study.
  Pimenta Amaral TM1, Campos CC, Moreira dos Santos TP, Leles CR, Teixeira AL, Teixeira MM, Bittencourt H, Silva TA.